CLINICAL TRIAL: NCT01248845
Title: Comparative Effects on Diaphragmatic Electrical Activity and Respiratory Pattern of Various Levels of Assistance in Pressure Support and in Neurally Adjusted Ventilatory Assist
Brief Title: Comparative Effects on Diaphragmatic Electrical Activity and Respiratory Pattern of Various Levels of Assistance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties to enroll patients
Sponsor: Prof. Philippe Jolliet (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Sponsor-Investigator, Prof. Philippe Jolliet, Main investigator, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: EMG_titr
Record Dates: First submitted 2010-08-20; First posted 2010-11-25 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Failure
Keywords: Mechanical ventilation; Electrical diaphragmatic activity
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Titration of various level of assistance — Exploration of the effects on diaphragmatic electrical activity (EMG) and on respiratory pattern of various level of assistance delivered by the ventilator in intubated spontaneously breathing patients in pressure support (PS) and in Neurally Adjusted Ventilatory Assist (NAVA) by step by step increasing of the level of assistance. Flow, airway pressure, transesophageal EMG signal and transcutaneous EMG signal will be recorded.

SUMMARY:
Exploration of the effects on diaphragmatic electrical activity (EMG) and on respiratory pattern of various level of assistance delivered by the ventilator in intubated spontaneously breathing patients in pressure support (PS) and in Neurally Adjusted Ventilatory Assist (NAVA) by step by step increasing of the level of assistance. Flow, airway pressure, transesophageal EMG signal and transcutaneous EMG signal will be recorded.

DETAILED DESCRIPTION:
Exploration of the effects on diaphragmatic electrical activity (EMG) and on respiratory pattern of various level of assistance delivered by the ventilator in intubated spontaneously breathing patients in pressure support (PS) and in Neurally Adjusted Ventilatory Assist (NAVA) by step by step increasing of the level of assistance. Flow, airway pressure, transesophageal EMG signal and transcutaneous EMG signal will be recorded.

Aims of the study:

1. To study the electrical diaphragmatic signal variations and the ventilatory profile variations under various level of assistance (delivered by the ventilator) in PS and in NAVA in intubated spontaneously breathing patients
2. To compare a non invasive technique of diaphragmatic electrical activity recording under various levels of assistance with the invasive reference technique

ELIGIBILITY:
Inclusion Criteria:

- Patients admitted to the ICU, intubated for acute respiratory failure, and ventilated in PS mode will be eligible for inclusion in the study.

Exclusion Criteria:

* Severe hypoxemia requiring an FIO2 > 0.5
* hemodynamic instability (defined as the need for high doses of catecholamines namely ≥ 0.5 μg/kg min- and/or high need in volume resuscitation namely more than two litres of crystalloids in two hours-)
* oesophageal problem such as hiatal hernia, oesophageal varicosities, oesophageal surgery;
* active upper gastro-intestinal bleeding;
* known coagulation disorder;
* any other contraindication to the insertion of a naso-gastric tube;
* poor short term prognosis (death expected within the next seven days)
* age < 18 years old.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Electrical diaphragmatic signal variations and ventilatory profile variations under various level of assistance
  To study the electrical diaphragmatic signal variations and the ventilatory profile variations under various level of assistance (delivered by the ventilator) in Pressure and in Neurally adjusted ventilatory assist in intubated spontaneously breathing patients

SECONDARY OUTCOMES:
Compare a non invasive technique of diaphragmatic electrical activity recording under various levels of assistance with the invasive reference technique.
  To compare a non invasive technique of diaphragmatic electrical activity recording under various levels of assistance with the invasive reference technique.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Jolliet, Professor, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- CHUV, University hospital of lausanne, Lausanne, Switzerland